CLINICAL TRIAL: NCT07000058
Title: Wide-Awake Local Anesthesia No Tourniquet (WALANT) With Versus Without Hyaluronidase for Hand Surgery
Status: Active, not recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Misr University for Science and Technology (Other)
Responsible Party: Principal Investigator, Emad Lotfy Mohammed Ahmed, Lecturer of anesthesia& pain, Misr University for Science and Technology
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2022/0103
Record Dates: First submitted 2025-05-23; First posted 2025-05-31 (Actual); Last update posted 2025-07-29 (Actual); Status verified 2025-07

CONDITIONS: Hand Surgery; Local Infiltration
Keywords: WALANT; Wide-Awake; Hand surgery; Hyaluronidase
MeSH Terms: interventions — Hyaluronoglucosaminidase; Lidocaine

STUDY DESIGN:
Intervention Model Description: Two groups of participants will receive WALANT technique;
  1. Group A (n=50); WALANT with Hyaluronidase
  2. Group B (n=50); WALANT without Hyaluronidase
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: All the above selected are blind regarding the used technique of anesthesia
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (n=50): WALANT with Hyaluronidase (Experimental): Patients received a mixture of hyaluronidase 15 IU to every 1 ml lidocaine 1% mixture (a solution composed of epinephrine 1:200,000 and lidocaine 1%). Buffered to reduce injection pain by 1 ml of sodium bicarbonate 8.4% for every 10 ml of the local anesthetic mixture.
  Interventions: Drug: Hyaluronidase and Lidocaine 1% mixture
- Group B (n=50): WALANT without Hyaluronidase: (Active Comparator): A mixture of epinephrine 1:200,000 and lidocaine 1% buffered to reduce injection pain by 1 ml of sodium bicarbonate 8.4% for every 10 ml of the local anesthetic mixture.
  Interventions: Drug: lidocaine 1 % mixture

INTERVENTIONS:
Drug: Hyaluronidase and Lidocaine 1% mixture — in group A hyaluronidase is expected to shorten the onset of action and prolong the duration of action of lidocaine 1% mixture than in group B where lidocaine 1% mixture only will be given
  Other Names: Hyalase
  Arms: Group A (n=50): WALANT with Hyaluronidase
Drug: lidocaine 1 % mixture — lidocaine 1 % mixture includes; A mixture of ( epinephrine 1:200,000 and lidocaine 1% ) buffered by 1 ml of sodium bicarbonate 8.4% for every 10 ml of the local anesthetic mixture.
  Other Names: Xylocaine 1%
  Arms: Group B (n=50): WALANT without Hyaluronidase:

SUMMARY:
The WALANT (Wide Awake Local Anesthesia No Tourniquet) method, introduced by Dr. Donald H. Lalonde over a decade ago, has gained popularity due to its favorable outcomes and patient satisfaction. This technique involves injecting diluted lidocaine and epinephrine, which helps control pain and bleeding without the discomfort of a tourniquet.

This research will explore the use of hyaluronidase to enhance the WALANT technique. The study hypothesize that adding hyaluronidase would improve the onset speed and duration of pain control. A double-blinded study involving 100 patients compared WALANT with hyaluronidase (Group A) to WALANT without Hyaluronidase (Group B).

DETAILED DESCRIPTION:
Background: Hand surgery, being one of the most frequent outpatient procedures, remains undecided regarding the ideal anesthesia technique. Wide-Awake Local Anesthesia No Tourniquet (WALANT) is one of the frequently used anesthesia techniques by some hand surgeons (8%).

Objective: The study aims to evaluate the impact of hyaluronidase administration on the onset and persistence of WALANT in hand surgery.

Patients and Methods: This Prospective, randomized, double-blind clinical trial will be conducted in Souad Kafafi University Hospital (SKUH), faculty of medicine, Misr University for Science and Technology (MUST).

One hundred patients (18-60years old) with ASA class I or II who will be scheduled for hand surgery. They will be equally divided into two groups: Group A (n =50) WALANT with hyaluronidase technique: Patients will receive a mixture of hyaluronidase 15 IU to every 1 ml lidocaine 1% mixture. Group B (n =50) WALANT without hyaluronidase technique: Patients will receive a mixture of lidocaine 1%. The infiltrative local anesthesia will be administered at the appropriate site in subcutaneous tissue just deep to the incisional site to produce tumescent local anesthesia. The onset time and duration of postoperative analgesia will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* One hundred individuals scheduled for hand surgery
* between the ages of 18 and 60 years old,
* of both sexes
* American Society of Anesthesiologists (ASA) classification I or II.
* were randomized 1:1 to either Group A; (Receiving WALANT with hyaluronidase) or Group B; (Receiving WALANT without hyaluronidase).

Exclusion Criteria:

* Pregnant women,
* patients who refused the terms of the research consent statement,
* psychiatric illness,
* uncooperative patient,
* patients with history of allergy to local anesthetic drugs,
* cardiac arrhythmia,
* patients with bleeding tendency,
* patients with low flow finger perfusion state such as Burger disease and Raynaud's disease,
* patients with connective tissue disease such as Scleroderma
* suspicious disease with malignancy and hand infection

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-06-20 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Onset time of analgesia. | from time of drug injection to start time of analgesia
  time to start analgesia

SECONDARY OUTCOMES:
Duration of postoperative analgesia | from onset time of analgesia to end of analgesia time postoperatively
  duration of analgesia
Pain intensity | from start of pain postoperatively till the end of first 24 hours postoperatively
  Pain intensity measured by Numerical Rating Scale (NRS)
The amount of morphine used | From start of postoperative pain to end of first 24 hours postoperatively
  Dose of morphine used for analgesia postoperatively
Amount of bleeding | From start of surgery to end of sugery
  Volume of blood loss
Patient satisfaction | From start of anesthesia till the end of first 24 hours postoperatively
  Patient comfort with the technique

CONTACTS AND LOCATIONS:
Overall Officials: Mohammed Hani Kamal, Prof., Study Chair — Anesth.&pain; Mohammed Safwat Hamza, Ass. prof., Study Director — Orthopedics
Locations (1):
- Misr University for Science and Technology, Giza, Giza Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Demographic Information: Age, sex, race, and other relevant demographic details.
  Baseline Characteristics: Health status, medical history, and any pre-existing conditions prior to the trial.
  Treatment Assignment: Information on the intervention or treatment each participant received.
  Outcome Measures: Data on primary and secondary outcomes as defined in the trial protocol.
  Adverse Events: Reports of any side effects or adverse events experienced by participants during the trial.
  Follow-up Data: Information collected during follow-up periods, including long-term outcomes.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: After 5 months from today and wil be available for one year
Access Criteria: Researchers:
  Who: Academic researchers, industry scientists, and regulatory agencies. What: Full IPD, including demographic data, treatment assignments, and outcome measures.
  How: Through data sharing platforms or repositories after submitting a research proposal and obtaining necessary approvals.
  Regulatory Authorities:
  Who: Agencies like the FDA or EMA. What: Full IPD and supporting documentation for oversight and review. How: Direct access during the review process of clinical trial applications.
  Data Sharing Initiatives:
  Who: Collaborating institutions and consortia. What: Aggregated or anonymized IPD for meta-analyses or systematic reviews. How: Via established partnerships and shared databases.
  Public and Patient Advocacy Groups:
  Who: Organizations seeking to promote transparency. What: Summary data and aggregated results, but not individual-level data. How: Through publicly available reports or dashboards.

REFERENCES:
- [Background] Farzam R, Deilami M, Jalili S, Kamali K. Comparison of Anesthesia Results between Wide Awake Local Anesthesia no Tourniquet (WALANT) and Forearm Tourniquet Bier Block in Hand Surgeries: A Randomized Clinical Trial. Arch Bone Jt Surg. 2021 Jan;9(1):116-121. doi: 10.22038/abjs.2020.49526.2487. PMID 33778124
- [Background] O'Neill N, Abdall-Razak A, Norton E, Kumar A, Shah H, Khatkar H, Alsafi Z, Agha R. Use of Wide-Awake Local Anaesthetic No Tourniquet (WALANT) in upper limb and hand surgery: A systematic review protocol. Int J Surg Protoc. 2020 Mar 13;20:8-12. doi: 10.1016/j.isjp.2020.03.001. eCollection 2020. PMID 32258835
- [Background] Seretis K, Boptsi A, Boptsi E, Lykoudis EG. The Efficacy of Wide-Awake Local Anesthesia No Tourniquet (WALANT) in Common Plastic Surgery Operations Performed on the Upper Limbs: A Case-Control Study. Life (Basel). 2023 Feb 4;13(2):442. doi: 10.3390/life13020442. PMID 36836799